CLINICAL TRIAL: NCT05781269
Title: Metabolic Syndrome and Severe Obesity: Randomized Nutritional Trial to Study Long Term Effect of Very-low-calories Ketogenic Diet (VLCKD) on Weight Control and Cardiovascular Risk Factors
Brief Title: Long Term Effect of Very-low-calories Ketogenic Diet on Weight Control and Cardiovascular Brisk Factors (KETOHEART)
Acronym: KETOHEART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43J001
Record Dates: First submitted 2023-02-26; First posted 2023-03-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Morbid Obesity
Keywords: VLCKD; obesity; metabolic syndrome; cardiovascular risk
MeSH Terms: conditions — Obesity; Obesity, Morbid; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLCKD-group (Experimental): The VLCKD will be applied with the specific products of the ketogenic protocol supplied by Laboratoire Therascience starting from the Active Phase. During this phase the patients will take 4-6 LIGNAFORM products which will be followed by the Selective Phase in which in one or both of the main meals the LIGNAFORM product will be replaced with a protein dish and the phases of reintroduction of fruit (phase three), dairy products and legumes (phase four), bread and derivatives (phase five) and cereals (phase 6). At the end of the previous phases, a normocaloric maintenance diet will be set, with a carbohydrate intake not exceeding 45% of total daily calories. In these subjects, VLCKD diet will be maintained for 2 weeks every 2 months of maintenance diet.
  Interventions: Other: VLCKD
- r-MedDiet (Experimental): The dietary treatment of the r-MedDiet group will provide for an average caloric deficit equal to 1000 kcal of the estimated total daily energy expenditure starting from the basal metabolic rate measured with indirect calorimetry and multiplied by the level of physical activity (LAF) defined on the basis of the Godin questionnaire. The diet will be personalized in 3 or 5 meals/day. Upon reaching the target weight, a Mediterranean-type diet plan will be set with a caloric intake equal to the estimated energy requirement
  Interventions: Other: r-MedDiet

INTERVENTIONS:
Other: VLCKD — VLCKD diet treatment with medical food
  Arms: VLCKD-group
Other: r-MedDiet — Mediterranean diet treatment
  Arms: r-MedDiet

SUMMARY:
The growing obesity pandemic has a major impact on global cardiovascular (CVD)-related morbidity and premature mortality, severely compromising the quality of life of those affected and significantly increasing costs for the healthcare system.

Numerous scientific evidences have demonstrated that a moderate weight loss (5-10% of the initial body weight) is already sufficient to determine the improvement of the cardiometabolic risk factors associated with overweight and obesity. With a view to obtaining a more significant weight loss in the initial stages of dietary treatment, in the last 10 years, the very low-calorie ketogenic diet (VLCKD) has become a strategy for the treatment of obesity and its comorbidities, also allowing to limit therapeutic failure and the high drop-out typical of traditional low-calorie diets.

The present study aims to study the long-term efficacy (36 months) of VLCKD in patients with severe obesity and metabolic syndrome, on weight loss, on single factors of the metabolic syndrome compared to a restrictive Mediterranean diet.

One hundred subjects with severe obesity and metabolic syndrome will be recruited and randomly assigned to VLCKD or to restrictive Mediterranean diet. Anthropometric parameters, metabolic status blood pressure, degree of arterial stiffness, prevalence and severity of snoring and OSA, cardiac systolic and diastolic function, the autonomic nervous control mode of the circulation will be evaluated at baseline, after one month and at the end of the study.

DETAILED DESCRIPTION:
The present study aims to study the long-term efficacy (36 months) of VLCKD in patients with severe obesity and metabolic syndrome, on weight loss, on single factors of the metabolic syndrome, on the plasma concentration of specific adipokines and myokines on the properties of arterial wall, cardiovascular function, and sleep quantity and quality compared to a restrictive Mediterranean diet.

The studied population includes men and women between the ages of 55 and 75, with no documented history of CVD, severely obese (BMI ≥30 e <50 kg / m2) and at least three positive factors for metabolic syndrome. The patient, after consideration of inclusion and exclusion factors, are enrolled for 36 months and randomly divided into two groups (50 patients for group): group 1 is assigned to VLCKD diet treatment with medical food (VLCKD-group) whereas group 2 followed Mediterranean diet treatment (r-MedDiet). Medical Foods products are provided by Therascience. For both groups, the achievement of the objective is set as a variation of 20% compared to the initial weight. Throughout the study, the long-term efficacy of VLCKD compared with a restrictive Mediterranean diet will be evaluated on the modification of anthropometric parameters (weight, waist circumference, hip circumference, impedance test) metabolic status (using blood chemistry tests for the evaluation of Blood glucose, glycosylated hemoglobin, insulin, total cholesterol, HDL, triglycerides, adiponectin and irisin), blood pressure (by sphygmomanometer), degree of arterial stiffness (by Pulse Wave Velocity carotid-femoral), prevalence and severity of snoring and OSA (by polysomnography), cardiac systolic and diastolic function (by three-dimensional echocardiography), the autonomic nervous control mode of the circulation (by analysis HRV, Arterial Baroreflex Sensitivity). .

These evaluations will be carried out at pre-established and different times (T0-T22) during the entire duration of the study.

The dietary treatment of the r-MedDiet group will provide for an average caloric deficit equal to 1000 kcal of the estimated total daily energy expenditure starting from the basal metabolic rate measured with indirect calorimetry and multiplied by the level of physical activity (LAF) defined on the basis of the Godin questionnaire. The diet will be personalized in 3 or 5 meals/day. Upon reaching the target weight, a Mediterranean-type diet plan will be set with a caloric intake equal to the estimated energy requirement. The VLCKD will be applied with the specific products of the ketogenic protocol supplied by Laboratoire Therascience starting from the Active Phase. During this phase the patients will take 4-6 LIGNAFORM products which will be followed by the Selective Phase in which in one or both of the main meals the LIGNAFORM product will be replaced with a protein dish and the phases of reintroduction of fruit (phase three), dairy products and legumes (phase four), bread and derivatives (phase five) and cereals (phase 6). At the end of the previous phases, a normocaloric maintenance diet will be set, with a carbohydrate intake not exceeding 45% of total daily calories. In these subjects, VLCKD diet will be maintained for 2 weeks every 2 months of maintenance diet.

ELIGIBILITY:
Inclusion Criteria:

* Men between the ages of 55 and 75 with no documented history of CVD (except NYHA class I and II heart failure or valvular heart disease)
* Women aged 60 to 75, with no documented history of CVD (except NYHA class I and II heart failure or valvular heart disease)
* BMI ≥30 and <50kg/m2-At least three positive factors for metabolic syndrome according to the harmonized definition (IDF --------2009)
* Availability to be followed in the follow-up at the San Michele Hospital IRCCS Istituto Auxologico Italiano in Milan

Exclusion Criteria:

* Long QT >0.44 s, known arrhythmia, cardiomyopathy, heart failure (NYHA classes III-IV)
* Hypokalemia, hypernatremia
* Persistent diarrhea
* Acidosis (metabolic or respiratory) even if compensated
* Acute heart failure, transient ischemic attack or stroke in the previous 12 months
* Pregnancy or breastfeeding
* chronic renal insufficiency (creatinine >1.5 and/or creatinine clearance <45 mL/min), history -positive for previous episodes of acute renal failure
* Autoimmune diseases (TCA relative contraindication)
* History of previous pancreatitis
* Symptomatic cholelithiasis
* Hepatic insufficiency and/or ALT and AST > 3 times the upper limit
* Stubborn constipation or history of intestinal occlusions/subocclusions
* Type 1 diabetes
* History of previous cancer within the first 5 years of follow-up
* Active eating disorder or history of bulimia and anorexia nervosa, active severe binge eating,
* Psychiatric disorders not in compensation or at risk of decompensation
* Alcoholism, substance abuse
* Ongoing pharmacological therapy with topiramate, zonisamide, acetazolamide, valproic acid- - ----- - chronic therapy with diuretics (which cannot be suspended even temporarily), SGLT2 -inhibitors (due to the risk of euglycemic diabetic ketoacidosis) and beta blockers.
* Known primary pathologies of carnitine metabolism or beta oxidation

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline body weight at 36 months | baseline, 36 month
  body weight measured to the nearest 0.1 Kg with a calibrated weight scale
change from baseline fasting glucose in mg/dl at 36 months | baseline, 36 month
  blood chemistry tests for the evaluation of blood glucose
change from baseline HDL cholesterol, triglycerides at 36 months | baseline, 36 month
  blood chemistry tests for the evaluation of HDL cholesterol, triglycerides
change from baseline blood pressure in mmHg at 36 months | baseline, 36 months
  measurement of systolic and diastolic pressure using using an aneroid sphygmomanometer with the appropriate cuff
change from baseline distensibility of the carotid, radial and femoral arteries in m/s at 36 months | baseline, 36 months
  arterial stiffness measured by Pulse Wave Velocity carotid-femoral
change from baseline waist circumference in cm at 36 months | baseline, 36 months
  waist circumference using a non-stretch tape to the nearest 0.5 cm

SECONDARY OUTCOMES:
change from baseline total and LDL cholesterol in mg/dl at 36 months | baseline, 36 months
  blood chemistry tests for the evaluation of total cholesterol, LDL cholesterol
change from baseline % of subjects with obstructive sleep apnea at 36 months | baseline, 36 months
  apnea hypopnea index using polysomnography
change from baseline cardiac systolic and diastolic function at 36 months | baseline, 36 months
  evaluation of the cardiac systolic and diastolic function using by three-dimensional echocardiography
change from baseline autonomic nervous control mode of the circulation at 36 months | baseline, 36 months
  by analysis HRV, Arterial Baroreflex Sensitivity
change from baseline insulin in mU/ml at 36 month | baseline, 36 months
  blood chemistry tests for the evaluation of insulin
change from baseline glycated hemoglobin in mmol/mol at 36 month | baseline, 36 months
  blood chemistry tests for the evaluation of glycated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bertoli, MD, Study Chair — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

REFERENCES:
- [Background] Zomer E, Gurusamy K, Leach R, Trimmer C, Lobstein T, Morris S, James WP, Finer N. Interventions that cause weight loss and the impact on cardiovascular risk factors: a systematic review and meta-analysis. Obes Rev. 2016 Oct;17(10):1001-11. doi: 10.1111/obr.12433. Epub 2016 Jun 21. PMID 27324830
- [Background] Diabetes Prevention Program Research Group; Knowler WC, Fowler SE, Hamman RF, Christophi CA, Hoffman HJ, Brenneman AT, Brown-Friday JO, Goldberg R, Venditti E, Nathan DM. 10-year follow-up of diabetes incidence and weight loss in the Diabetes Prevention Program Outcomes Study. Lancet. 2009 Nov 14;374(9702):1677-86. doi: 10.1016/S0140-6736(09)61457-4. Epub 2009 Oct 29. PMID 19878986
- [Background] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- [Background] Wing RR, Lang W, Wadden TA, Safford M, Knowler WC, Bertoni AG, Hill JO, Brancati FL, Peters A, Wagenknecht L; Look AHEAD Research Group. Benefits of modest weight loss in improving cardiovascular risk factors in overweight and obese individuals with type 2 diabetes. Diabetes Care. 2011 Jul;34(7):1481-6. doi: 10.2337/dc10-2415. Epub 2011 May 18. PMID 21593294
- [Background] Caprio M, Infante M, Moriconi E, Armani A, Fabbri A, Mantovani G, Mariani S, Lubrano C, Poggiogalle E, Migliaccio S, Donini LM, Basciani S, Cignarelli A, Conte E, Ceccarini G, Bogazzi F, Cimino L, Condorelli RA, La Vignera S, Calogero AE, Gambineri A, Vignozzi L, Prodam F, Aimaretti G, Linsalata G, Buralli S, Monzani F, Aversa A, Vettor R, Santini F, Vitti P, Gnessi L, Pagotto U, Giorgino F, Colao A, Lenzi A; Cardiovascular Endocrinology Club of the Italian Society of Endocrinology. Very-low-calorie ketogenic diet (VLCKD) in the management of metabolic diseases: systematic review and consensus statement from the Italian Society of Endocrinology (SIE). J Endocrinol Invest. 2019 Nov;42(11):1365-1386. doi: 10.1007/s40618-019-01061-2. Epub 2019 May 20. PMID 31111407
- [Background] Esposito K, Kastorini CM, Panagiotakos DB, Giugliano D. Mediterranean diet and weight loss: meta-analysis of randomized controlled trials. Metab Syndr Relat Disord. 2011 Feb;9(1):1-12. doi: 10.1089/met.2010.0031. Epub 2010 Oct 25. PMID 20973675